CLINICAL TRIAL: NCT05449548
Title: Lenalidomide in the Treatment of Mucosal Behçet's Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: lenalidomide in BS
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-06

CONDITIONS: Oral Ulcer
MeSH Terms: conditions — Oral Ulcer | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention with lenalidomide (Experimental): All subjects will be treated with lenalidomide 10mg/day.
  Interventions: Drug: Lenalidomide 10 mg

INTERVENTIONS:
Drug: Lenalidomide 10 mg — All subjects will be treated with lenalidomide 10mg/day with a regular follow-up of 12 weeks, followed by a 4-week observation after cessation of lenalidomide.
  Other Names: Lenalidomide

SUMMARY:
The study is to evaluate the efficacy and safety of lenalidomide in the treatment of oral ulcers in adult patients with refractory mucosal Behcet's syndrome.

DETAILED DESCRIPTION:
Behçet's Syndrome (BS) is a systemic vasculitis involving blood vessels of all sizes. It is characterised by recurrent oral and genital ulcers, skin lesions, musculoskeletal, ophthalmic, large vessel and intestinal involvements. Mucosal BS is the most common phenotype of BS, commonly treated with thalidomide and colchicine, yet some patients respond poorly or had limited use due to side effects.

Lenalidomide, a second-generation derivative of thalidomide, has a role as an angiogenesis inhibitor, an antineoplastic agent and an immunomodulator.

Its neurotoxicity and reproductive toxicity are significantly reduced, and the ability of TNF-alpha inhibition is significantly increased.

Reports on lenalidomide for refractory mucosal BS have been mostly case reports and preliminary studies, clinical trials are lacking.

This is a single-centre, prospective, open-label, single-arm study to evaluate the efficacy and safety of lenalidomide in the treatment of refractory mucosal BS; with the rate of complete remission of oral ulcers in subjects at 12 weeks as the primary endpoint; partial remission of oral and genital ulcers, non-response rate and BS disease activity as secondary endpoints; and adverse events and newly-developed BS-related symptoms as safety endpoints.

This study aims to enroll adult patients with refractory mucosal BS with a stable dosage of low-dose glucocorticoids and/or other conventional immunomodulators. All subjects will be treated with lenalidomide 10mg/day with regular follow-up, those having adverse effects will be evaluated by investigators and adjusted to 5mg/day if necessary, with glucocorticoids and immunosuppressive agents adjusted as needed. Each subject will complete a 12-week treatment period, followed by 4 weeks of observation after cessation of lenalidomide.

ELIGIBILITY:
Inclusion Criteria:

* Patients that can understand and voluntarily sign an informed consent document prior to the study;
* Male and female subjects ≥ 18 years and ≤ 65 years of age at the time of signing the informed consent document.
* Fulfilling the ICBD (International Conference on Behcet's Disease) criteria(2013);
* Presented with active mucosal lesions: Subjects must have at least 1 oral ulcer within 4 weeks after the screening visit and at least 2 oral ulcers on the day of enrollment; subjects may be with or without genital ulcers and (or) skin lesions.
* Refractory mucosal lesions: Subjects must experience at least 2 relapses of oral ulcers during 3 consecutive months of conventional treatment with corticosteroids and(or) immunosuppressants.
* Without major organ involvement, including active gastrointestinal, ocular, nervous system, and major vessel involvement; previous major organ involvement is allowed if it occurred at least 1 year prior to the screening visit and is not active at the time of enrollment.; subjects with arthritis are permitted.

Exclusion Criteria: The presence of any of the following will exclude a subject from the study enrollment.

Exclusion Criteria:

* Pregnant women or breastfeeding mothers, Male and female patients with recent fertility requirements.
* Skin and mucosal lesions should exclude erythema multiforme, syphilis, Sweet disease, Stevens-Johnson syndrome, acne vulgaris, herpes simplex infection, periodic granulocytopenia, and acquired immunodeficiency.
* Subjects with Behçet's syndrome-related active major organ involvement that requires aggressive immunosuppressive therapy, including active gastrointestinal, ocular, nervous system, and major vessel involvement.
* Severe Concomitant disease: including heart failure(≥level Ⅲ, NYHA), respiratory failure, renal insufficiency (Serum creatinine ≥ 1.5 mg/dL ), hepatic insufficiency(Aspartate transaminase (AST) and alanine transaminase (ALT) ≥ 2 X ULN.), myelosuppression(WBC<3.0×109/L or N<1.5×109/L, HGB≤85g/L, PLT<100×109/L), peripheral neuropathy.
* Acute severe infections such as sepsis and cellulitis, active hepatitis B or C virus infection, active tuberculosis, and history of a positive test for, or any clinical suspicion of, human immunodeficiency virus (HIV).
* Patients with malignancy, or any history of malignancy within the 5 years prior to the screening phase, risk factors for myocardial infarction (including a history of thrombosis), or hypercoagulability.
* History of use of lenalidomide or thalidomide within 1 month before enrollment.
* Patients with allergies or contraindications to lenalidomide or thalidomide.
* Having received concomitant immune-modulating therapy or small molecule drugs. At least 5 terminal half-lives for all biologics, including, but not limited to, those listed below; within:

Ten days prior to the day of enrollment for tofacitinib and baricitinib Four weeks prior to the day of enrollment for etanercept Eight weeks prior to the day of enrollment for infliximab Ten weeks prior to the day of enrollment for adalimumab, golimumab, certolizumab, abatacept, and tocilizumab Six months prior to the day of enrollment for secukinumab

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The complete remission rate of oral ulcers in subjects after 12 weeks of treatment | 12 weeks
  A complete remission at week 12 was defined as participants who were oral ulcer-free at week 12.

SECONDARY OUTCOMES:
Percentage of participants who had an partial response of oral ulcer at Week 12 | 12 weeks
  A partial response at week 12 was defined as participants with a 50% or more reduction in the number of oral ulcers at week 12
Percentage of participants who had no response of oral ulcer at Week 12 | 12 weeks
  No response at week 12 was defined as all other participants at week 12
Percentage of participants who had a complete response of genital ulcer at Week 12 | 12 weeks
  A complete remission at week 12 was defined as participants who were genital ulcer-free at week 12.
Percentage of participants who had an partial response of genital ulcer at Week 12 | 12 weeks
  A partial response at week 12 was defined as participants with a 50% or more reduction in the number of genital ulcers at week 12
Percentage of participants who had no response of genital ulcer at Week 12 | 12 weeks
  No response at week 12 was defined as all other participants at week 12
Change from baseline on oral ulcer pain as measured by visual analogue scale (VAS) at week 12 | Baseline to week 12
  Pain of oral ulcers was measured using a 100 mm VAS scale. The participant was asked to draw a single line perpendicular to the VAS line at the point that represented the severity of their pain during the previous week, with 0 mm (the left-hand end of the scale) representing no pain and 100 mm (the right-hand end of the scale) representing the worst pain imaginable. The distance of the perpendicular line from the left-hand end of the scale was recorded.
  A negative change from baseline indicates improvement.
Change from baseline on genital ulcer pain as measured by visual analogue scale (VAS) at week 12 | Baseline to week 12
  Pain of genital ulcers was measured using a 100 mm VAS scale. The participant was asked to draw a single line perpendicular to the VAS line at the point that represented the severity of their pain during the previous week, with 0 mm (the left-hand end of the scale) representing no pain and 100 mm (the right-hand end of the scale) representing the worst pain imaginable. The distance of the perpendicular line from the left-hand end of the scale was recorded.
  A negative change from baseline indicates improvement.
Change from baseline in disease activity as measured by Behçet's Disease Current Activity Form (BDCAF) | Baseline to week 12
  The Behçet's Disease Current Activity Form (BDCAF) consists of 3 component scores: the Behçet's Disease Current Activity Index (BDCAI) score, the Patient's Perception of Disease Activity, and the Clinician's Overall Perception of Disease Activity.
  The BDCAI consists of 12 questions regarding disease manifestations over the previous 4 weeks, The score is the sum score of 12 items and ranges from 0 to 12. A higher score indicates a higher level of disease activity, and a negative change from baseline indicates improvement.
  The Patient's Perception of Disease Activity was assessed on a scale from 1 to 7, and the Clinician's Overall Perception of Disease Activity was assessed on a scale from 1 to 7. A higher score indicates a higher level of disease activity and a negative change from baseline indicates improvement.
Change from baseline in disease activity as measured by Behçet's Syndrome Activity Score (BSAS) at Week 12 | Baseline to week 12
  The Behçet's Syndrome Activity Score (BSAS) contains 10 questions that assess the number of new oral and genital ulcers and skin lesions, GI, CNS, vascular, and ocular involvement, and the participant's current level of discomfort. The Behçet's Syndrome Activity Score ranges from 0 to 100, with a higher score indicating a higher level of disease activity. A negative change from baseline indicates improvement.
Change from baseline in Behçet's Disease Quality of Life (BD Qol) Scores at week 12 | Baseline to week 12
  The Behçet's Disease Quality of Life questionnaire was developed to measure the influence of BD on a particpant's life. It consists of 30 self-completed itemized questions that measure disease- related restrictions on the participant's activities and their emotional response to these restrictions. The total score is the sum of all 30 items (each yes scores 1 and each no scores 0), with 0 representing no influence of Behçet's disease on a participant's quality of life and 30 representing the most severe influence. A negative change from baseline indicates improvement.
Change From baseline in Short Form-36 Health Status Questionnaire(SF-36) | Baseline to week 12
  Short Form-36 Health Status Questionnaire(SF-36) is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Corticosteroid-tapering effects. | Baseline to week 12
  The dosage of glucocorticoids will be tapered tailored to the disease activity of each participant, and the change of dosage from baseline will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjie Zheng, M.D., Principal Investigator — Department of Rheumatology, Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No